CLINICAL TRIAL: NCT00316758
Title: A Multi-center, Open Label, Extension Study to Evaluate the Long-term Safety and Tolerability of GK Activator (2) in Type 2 Diabetic Patients From Studies BM18248 or BM18249
Brief Title: A Study to Evaluate the Long-Term Safety and Tolerability of GK Activator (2) in Patients With Type 2 Diabetes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NC19794
Record Dates: First submitted 2006-04-20; First posted 2006-04-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: GK Activator (2); Drug: Metformin

INTERVENTIONS:
Drug: GK Activator (2) — Escalating doses bid
Drug: Metformin — As prescribed, in patients who were in study BM18249

SUMMARY:
This study will evaluate the long-term safety and tolerability of GK Activator (2) at doses ranging from 25mg - 100mg po bid, administered alone or in combination with metformin, in patients with type 2 diabetes. Eligible patients will be those who have completed study BM18248 (GK Activator (2) monotherapy) or BM18249 (GK Activator (2) and metformin); they will continue on the same treatment regimen (mono or combination therapy) as they received in the initial study. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients who have completed studies BM18248 or BM18249;
* patients considered by the investigator to be suitable for long term treatment with GK Activator (2).

Exclusion Criteria:

* type 1 diabetes mellitus;
* women who are pregnant, breast-feeding or not using adequate contraceptive methods.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory parameters, ECG. | Throughout study

SECONDARY OUTCOMES:
Mean change from original baseline in HbA1c, FPG, lipid profile. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (53):
- United States (21):
  - Chula Vista, California
  - Los Angeles, California
  - Spring Valley, California
  - West Hills, California
  - Hollywood, Florida
  - Kissimmee, Florida
  - Atlanta, Georgia
  - Arkansas City, Kansas
  - Butte, Montana
  - Binghamton, New York
  - Fayetteville, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Springdale, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Beaver, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Memphis, Tennessee
  - Federal Way, Washington
  - Renton, Washington
- Australia (2):
  - Camperdown
  - Heidelberg
- Bulgaria (4):
  - Dimitrovgrad
  - Pleven
  - Rousse
  - Sofia
- Canada (3):
  - Vancouver, British Columbia
  - London, Ontario
  - Montreal, Quebec
- Zagreb, Croatia
- Germany (9):
  - Bammental
  - Berlin
  - Essen
  - Giessen
  - Görlitz
  - Hamburg
  - Künzing
  - Nuremberg
  - Tann
- Guatemala City, Guatemala
- Hungary (3):
  - Budapest
  - Győr
  - Kecskemét
- Mexico (4):
  - Chihuahua City
  - Cuernavaca
  - Durango
  - Mexico City
- Poland (5):
  - Bialystok
  - Gdansk
  - Gorzów
  - Krakow
  - Wroclaw